CLINICAL TRIAL: NCT05598671
Title: A Comparative Study of Retrograde Ureteral Catheter Insertion or Not in Percutaneous Nephrolithotomy
Brief Title: Percutaneous Nephrolithotomy Without a Ureteral Catheter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Li Mingyong, MD, Associate professor, The First Affiliated Hospital of University of South China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nhfy0520
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Nephrolithotomy Percutaneous; Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without reverse insertion of a ureteral catheter (Experimental): Percutaneous nephrolithotomy without reverse insertion of a ureteral catheter
  Interventions: Procedure: PCNL without reverse insertion of a ureteral catheter
- Conventional (No Intervention): Percutaneous nephrolithotomy with reverse insertion of a ureteral catheter

INTERVENTIONS:
Procedure: PCNL without reverse insertion of a ureteral catheter — The ureteral catheter was not retrograde inserted during PCNL
  Arms: without reverse insertion of a ureteral catheter

SUMMARY:
Conventional Percutaneous nephrolithotomy (PCNL) surgery requires the patient to first undergo retrograde transurethral ureteroscopic insertion of the ureteral catheter in the lithotomy position, and then change the patient to the prone position. However, repeated operation on the ureter can bring about immediate and long-term negative effects, such as ureteral false way formation, ureteral damage, perforation, avulsion, catheter insertion into the vena cava, pricking the kidney, increased postoperative pain, urinary extravasation, scar formation, and ureteral narrowing. The study planned to perform the operation in the prone position without reverse insertion of a ureteral catheter in the PCNL surgery.

DETAILED DESCRIPTION:
The purpose of this single-center, single-blind, randomized trial was to evaluate the safety and efficacy of PCNL without reverse insertion of a ureteral catheter. It is planned to start in November 2022 and is expected to end in November 2024. Based on inclusion and exclusion criteria, 200 subjects were expected to be recruited. In a parallel group design, subjects were randomly assigned to two groups: the experimental group received PCNL without reverse insertion of a ureteral catheter , and the control group received traditional PCNL. The primary end point of the study was the incidence of postoperative complications according to the modified Clavien-Dindo complication grading system. Secondary end points included Stone-free rate, operation time, length of hospital stay, and medical costs. Measurement data were expressed as mean ± standard deviation (X ± S), and Student's t-test was used for intergroup comparisons. The counting data were expressed as frequency and percentage, and the chi-squared or Fisher's exact probability test were used for intergroup comparisons. The rank-sum test was used for grade data. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

· Patients with upper urinary tract stones who were 18 years of age or older and eligible for PCNL surgery.

Exclusion Criteria:

* patients with infectious calculi confirmed by preoperative CT examination and blood biochemical indexes.
* Patients with severe cardiac and pulmonary insufficiency, coagulation dysfunction and other obvious surgical contraindications.
* Patients with previous history of PCNL surgery on the affected side or nephrotomy.
* Patients with indwelling double J tube or nephrostomy tube before operation.
* Patients with renal trauma or congenital anomalies of urinary system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of fever | From the day of surgery to the day of discharge, up to 2 weeks.
  Fever was defined as axillary temperature greater than 38.5 ° C.
White blood cell count change value | Day 2 before surgery、hour 3 after the surgery
  The change value of White blood cell count between preoperative and postoperative
Neutrophils granulocyte change value | Day 2 before surgery、hour 3 after the surgery
  The change value of Neutrophils granulocyte between preoperative and postoperative
Hemoglobin change value | Day 2 before surgery、hour 3 after the surgery
  The change value of Hemoglobin between preoperative and postoperative
Hematocrit change value | Day 2 before surgery、hour 3 after the surgery
  The change value of Hematocrit between preoperative and postoperative
Rate of renal subcapsular hematoma | Day 2 after the surgery
  The proportion of postoperative renal subcapsular hematoma in all patients
Serum creatinine change value | Day 2 before surgery、Hour 3 after the surgery
  The change value of Serum creatinine between preoperative and postoperative
visual analog scale (VAS)pain score | Hour 2 after the surgery
  0: no pain; Less than 3 points: mild pain, tolerable; 4 points to 6 points: the patient's pain and affect sleep, still tolerable; 7-10: Patients have increasing pain, pain is unbearable, affect appetite, affect sleep.
Rate of hydrothorax | Day 2 after the surgery
  Hydrothorax appeared on the surgical side.

SECONDARY OUTCOMES:
Stone free rate | Day 2 after the surgery
  Residual stone less than 4mm in diameter was considered to have been cleared.
Operation time | During the procedure
  Operation time was defined as the time required from the surgeon's handwashing to the completion of surgical incision suture
length of hospital stay | 2 weeks after surgery
  Length of hospital stay indicated the number of days between the operation date and discharge date
Medical costs | 2 weeks after surgery
  All medical expenses incurred to treat stones.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyong Li, MD., Study Director — the First Affiliated Hospital of the University of South China
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to other researchers after the study Report are published.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the study report was published,but the duration is uncertain.
Access Criteria: When proper editing or review requirements are met, the study data will be available from the study manager after the study is completed.